CLINICAL TRIAL: NCT00890916
Title: Hand Function for Tetraplegia Using a Wireless Neuroprosthesis
Brief Title: Hand Function for Tetraplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6027-R
Record Dates: First submitted 2009-04-27; First posted 2009-04-30 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Spinal Cord Injury; Tetraplegia
Keywords: spinal cord injury; neuroprosthesis; functional electrical stimulation; quadriplegia
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Neuroprosthesis System (Experimental): Receives implanted device for hand function.
  Interventions: Device: FIRSTHAND System

INTERVENTIONS:
Device: FIRSTHAND System — Implanted neuroprosthesis with myoelectric control and electrical stimulation of multiple channels.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of an implanted stimulator for providing hand function to individuals with cervical level spinal cord injury. The device stimulates the paralyzed muscles of the hand and forearm. The user of the device controls the stimulation by moving muscles that are not paralyzed, such as a wrist or neck muscle. The ability of the user to pick up and move objects, as well as perform various activities such as eating, drinking, and writing.

DETAILED DESCRIPTION:
The overall object of this research is to provide restored functional abilities to individuals with cervical-level spinal cord injury through the use of an advanced wireless myoelectrically controlled battery-powered implanted neuroprosthetic system known as the "FIRSTHAND" System. This restored function can enable the individual to achieve greater independence in activities of daily living and an improved quality of life. Electrical stimulation of paralyzed muscles will be used to generate functional movements. The movements will be controlled using myoelectric signals generated from muscles under the subject's voluntary control. The specific hypotheses of this study are: 1) at least 75% of all subjects will be able to manipulate at least one more object in the Grasp-Release Test when using the advanced neuroprosthesis compared to without the neuroprosthesis. 2) At least 75% of all subjects will demonstrate an increased level of independence in at least one functional activity when using the advanced neuroprosthesis. 3) At least 75% of all subjects will demonstrate an average neuroprosthesis usage of at least three days/week.

ELIGIBILITY:
Inclusion Criteria:

* cervical level spinal cord injury;
* complete paralysis of fingers and thumbs;
* voluntary shoulder motion;
* electrically excitable forearm and hand musculature

Exclusion Criteria:

* extreme contractures of the joints;
* skeletal immaturity;
* extensive denervation in the forearm and hand;
* poor surgical risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2015-11-01 (Actual); Study Completion 2021-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin L Kilgore, PhD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peckham PH, Kilgore KL. Challenges and opportunities in restoring function after paralysis. IEEE Trans Biomed Eng. 2013 Mar;60(3):602-9. doi: 10.1109/TBME.2013.2245128. Epub 2013 Mar 7. PMID 23481680
- [Result] Kilgore KL, Bryden A, Keith MW, Hoyen HA, Hart RL, Nemunaitis GA, Peckham PH. Evolution of Neuroprosthetic Approaches to Restoration of Upper Extremity Function in Spinal Cord Injury. Top Spinal Cord Inj Rehabil. 2018 Summer;24(3):252-264. doi: 10.1310/sci2403-252. PMID 29997428
- [Result] Kilgore KL, Hoyen HA, Bryden AM, Hart RL, Keith MW, Peckham PH. An implanted upper-extremity neuroprosthesis using myoelectric control. J Hand Surg Am. 2008 Apr;33(4):539-50. doi: 10.1016/j.jhsa.2008.01.007. PMID 18406958
- See also: Cleveland FES Center website - research into restoring movement using neuroprostheses — http://fescenter.org/index.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Note that the data from the first three (of 10) participants was published in the Journal of Hand Surgery (2008; 33(4):539-50).
Groups:
- Neuroprosthesis System: Subjects who have undergone implantation of the neuroprosthesis system known as the FIRSTHAND/IST-12 System.
Period: Rehab - Neuroprosthesis (NP) "On"
Arm/Group | Neuroprosthesis System
Started | 10 (First Implanted Stimulator-Telemeter (IST-12) Implant.)
Grasp Release Pre-Test "ON" (Grasp Release Pre-Test results - Neuroprosthesis turned on. See Peckham et al.,Arch PM&R,2001) | 10
Completed | 10
Not Completed | 0
Period: Rehab - NP "Off"
Arm/Group | Neuroprosthesis System
Started | 10
Grasp Release Pre-Test "OFF" | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: C5/C6 Spinal Cord Injury
Groups:
- Neuroprosthesis System: Receives implanted device for hand function.
  FIRSTHAND System: Implanted neuroprosthesis with myoelectric control and electrical stimulation of multiple channels. Also known as the "IST-12" System.
Arm/Group | Neuroprosthesis System
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Grasp-Release Test [Median (Full Range); unit: Number of Completions] — The Grasp and Release Test (GRT) [Wuolle, 1994; Smith et al., 1996; Carroll et al., 2000; Peckham, 2001; Taylor et al., 2002; Mulcahey et al., 2004], is a pick-and-place test requires the participant to unilaterally acquire, move, and release six objects varying in weight and size. The objects are: 1) a small peg, 2) a wooden cube, 3) a small juice can, 4) a videotape, 5) a paperweight and a simulated fork task. The number of objects that the participant can successfully manipulate are scored.
  Number of Completions | 2 [0 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Grasp Release Test - Test of Functional Ability to Pick up and Move Objects
Description: Grasp and Release Test (GRT) - The Grasp and Release Test (GRT) [Wuolle, 1994; Smith et al., 1996; Carroll et al., 2000; Taylor et al., 2002; Mulcahey et al., 2004], developed at the Cleveland FES Center, has been utilized by multiple centers to show improvements in hand function after implantation of a neuroprosthesis and tendon transfers [Peckham, 2001]. This pick-and-place test requires the participant to unilaterally acquire, move, and release six objects varying in weight and size. The objects are: 1) a small peg, 2) a wooden cube, 3) a small juice can, 4) a videotape, 5) a paperweight (~1000g) and a simulated fork task (spring-loaded plunger). The number of objects that the participant can successfully manipulate are scored. Success in manipulating each object in the GRT is defined as the ability to pick up and place the object at least once within 30 seconds.
Time Frame: 6-9 weeks
Measure: Median (Full Range); unit: Number of Completions
Groups:
- Neuroprosthesis System: Subjects with the implanted FIRSTHAND/IST-12 System.
Arm/Group | Neuroprosthesis System
Number analyzed (Participants) | 10
Number of Completions
  Rehab - NP "OFF" | 2 [0 to 4]
  Rehab - NP "ON" | 5.5 [5 to 6]

ADVERSE EVENTS:
Arm/Group | Neuroprosthesis System
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neuroprosthesis System (N=10)
Device Infection (Infections and infestations) | 2 (2) — Device infection of any implanted component requiring removal of some or all components of system.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes